CLINICAL TRIAL: NCT04322110
Title: Pilot Study Fatty Liver and Obesity: MR Fat Quantification and MR Elastography During a Very Low-calorie-ketogenic Diet (Pronokal Method®) Versus a Low Calorie Diet
Brief Title: MR Fat Quantification and Elastography During a Very Low-calorie-ketogenic Diet (Pronokal Method®) vs a Low Calorie Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protein Supplies SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNK-FATLIV-2016-04
Record Dates: First submitted 2020-03-13; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2016-05

CONDITIONS: Liver Fat
Keywords: Low-Calorie-Ketogenic diet; Low Calorie Diet; Pronokal Method®; Fat reduction
MeSH Terms: conditions — Fatty Liver | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLCK diet group (Experimental): Subjects undergoing treatment with weight loss program PronoKal Method
  Interventions: Other: PronoKal Method
- Control group (Active Comparator): Subjects undergoing treatment with low calorie diet
  Interventions: Other: Low calorie diet

INTERVENTIONS:
Other: PronoKal Method — Multidisciplinary program of weight loss based on diet (initially ketogenic diet), physical activity and emotional support
  Arms: VLCK diet group
Other: Low calorie diet — Balanced hypocaloric diet (caloric intake 10% below basal metabolic rate) accompanied by physical exercise.
  Arms: Control group

SUMMARY:
Prospective, multicenter, open-label, randomized and controlled study of the effects of weight loss and reduced visceral fat on non-alcoholic fat infiltration into liver after a very low calorie ketogenic diet (VLCK diet) (Pronokal® Method) versus a hypocaloric diet, with a 6-month follow-up.

DETAILED DESCRIPTION:
The investigators will include obese patients with BMI higher than 30 kg / m2 to follow a standardized multidisciplinary weight-loss program (PronoKal® Method), which consists of a very-low-calorie diet, into which natural foods are gradually reintroduced, accompanied by physical exercise and emotional support, versus hypocaloric diet.

The aim of this study are see the reduction of fatty liver, visceral fat and improvement of hepatic stiffness during the weight loss treatment.

Patients will be visited monthly and data will recorded on 4 occasions: pre-inclusion, initial visit, 2-months visit (end of ketosis) and 6-months visit.

Hepatic fatty infiltration and visceral fat will be scanned by MRI and hepatic stiffness will be assessed by MR Elastography at: baseline, 2 months and 6 months. Also will be recorded anthropometric data (weight, BMI, waist circumference) and complete blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, older than 18 years
* Obese patients with BMI equal or over 30kg/m2
* Patients who agree to participate and sign the Informed Consent

Exclusion Criteria:

* Pregnant or lactating women.
* Patients weighing over 140 kg (by limitation of the MRI device)
* Patients on anti-obesity drugs (eg, sibutramine, orlistat and liraglutide) or weight-interfering medications (eg, topiramate). In such cases a wash out period of 3 months is required.
* Patients with alcohol intake > 20 g/day in women and > 30 g/day in men.
* Patients with liver failure or with pathologies that may affect the liver
* Patients with other causes of liver steatosis: chronic viral hepatitis and/or drug intake (corticosteroids, estrogens, NSAIDs, calcium antagonists, amiodarone, tamoxifen, tetracyclines, chloroquine, antiretrovirals, perhexiline).
* Patients with eating disorders.
* Patients with any psychiatric disorder (eg schizophrenia, bipolar disorder, substance abuse, severe depression).
* Patients receiving dicumarinic anticoagulants (Sintrom®).
* Patients taking corticosteroids.
* Patients with severe kidney failure (gfr <30).
* Patients with type 1 and type 2 diabetes mellitus.
* Patients with hemopathies, including coagulation disorders
* Patients with cardiovascular or cerebrovascular disease (of heart rate disorders, recent infarction [<6m], unstable angina, decompensated heart failure, recent stroke [<6m]).
* Patients in acute attack of gout.
* Patients with renal lithiasis verified by ultrasound.
* Patients with cholelithiasis verified by ultrasound.
* Patients with electrolyte imbalance, according to medical criteria.
* Patients with orthostatic hypotension.
* Patients with cancer or history of cancer who have not been discharged from oncology
* Patients who are not expected to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Liver fatty infiltration at 6 months | 6 months
  Liver fatty infiltration percentage, measured by a MRI technique of fat liver quantification, fat at the end of treatment

SECONDARY OUTCOMES:
Liver fatty infiltration at 2 months | 2 months
  Liver fatty infiltration percentage, measured by a MRI technique of fat liver quantification, at the end of ketosis
Visceral fat at 2 months | 2 months
  Viceral fat measured by the area in squared centimeters at the level of the 3rd vertebrae, using MRI technique, at the end of ketosis.
Visceral fat at 6 months | 6 months
  Viceral fat measured by the area in squared centimeters at the level of the 3rd vertebrae, using MRI technique, at the end of treatment.
Liver stiffness at 2 months | 2 months
  Liver stiffness detected by MR Elastography at the end of ketosis
Liver stiffness at 6 months | 6 months
  Liver stiffness detected by MR Elastography at the end of treatment
Size of adrenal gland at 2 months | 2 months
  Linear size in centimetres of adrenal gland at the end of ketosis, measured by MRI.
Size of adrenal gland at 6 months | 6 months
  Linear size in centimetres of adrenal gland at the end of treatment, measured by MRI.
Body Weight loss at 2 months | 2 months
  Change in body weight from baseline to end of ketosis.
Body Weight loss at 6 months | 6 months
  Change in body weight from baseline to end of treatment.
Salivary cortisol levels at 2 months | 2 months
  Salivary cortisol levels at the end of ketosis
Salivary cortisol levels at 6 months | 6 months
  Salivary cortisol levels at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Walmir Coutinho, Ph, Principal Investigator — IEDE - Instituto Estadual de Diabetes e Endocrinologia; Guilherme Moura da Cunha, Ph, Principal Investigator — CDPI - Clínica de Diagnóstico por Imagen

REFERENCES:
- [Derived] Cunha GM, Guzman G, Correa De Mello LL, Trein B, Spina L, Bussade I, Marques Prata J, Sajoux I, Countinho W. Efficacy of a 2-Month Very Low-Calorie Ketogenic Diet (VLCKD) Compared to a Standard Low-Calorie Diet in Reducing Visceral and Liver Fat Accumulation in Patients With Obesity. Front Endocrinol (Lausanne). 2020 Sep 14;11:607. doi: 10.3389/fendo.2020.00607. eCollection 2020. PMID 33042004

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04322110/Prot_SAP_000.pdf